CLINICAL TRIAL: NCT03861156
Title: A Phase II Study to Assess the Safety and Efficacy of D-0316 in Patients With Locally Advanced/Metastatic Non Small Cell Lung Cancer Whose Tumors Are Epidermal Growth Factor Receptor Mutation Positive
Brief Title: D-0316 in Patients With EGFR Positive Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBIO-102
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumor; NSCLC; EGFR T790M

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-0316 (Experimental): Firstly, D-0316 was orally given 75mg for a cycle(21 days), if tolerated, the dose will be increased to 100mg. Otherwise, the dose will be maintained at 75mg.
  Interventions: Drug: D-0316

INTERVENTIONS:
Drug: D-0316 — Firstly, D-0316 was orally given 75mg for a cycle(21 days), if tolerated, the dose will be increased to 100mg. Otherwise, the dose will be maintained at 75mg.

SUMMARY:
A Phase II, Open Label, Single-arm Study to Assess the Safety and Efficacy of D-0316 in Patients with Locally Advanced/Metastatic Non Small Cell Lung Cancer whose Disease has Progressed with Previous Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and whose Tumours are Epidermal Growth Factor Receptor Mutation and T790M Mutation Positive

DETAILED DESCRIPTION:
This is a phase II, open label, single arm study assessing the safety and efficacy of D-0316 (Firstly, D-0316 was orally given 75mg for a cycle(21 days), if tolerated, the dose will be increased to 100mg. Otherwise, the dose will be maintained at 75mg.) in patients with a confirmed diagnosis of Epidermal Growth Factor Receptor mutation positive and T790M mutation positive NSCLC,who have progressed following prior therapy with an approved Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) agent. The primary objective of the study is to assess the efficacy of D-0316 by assessment of Objective Response Rate according to RECIST 1.1 by an Independent Central Review.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* Histologically or cytologically proven diagnosis of NSCLC that is locally advanced or metastatic.
* Radiological documentation of disease progression while on a previous continuous treatment with an first or second generation of EGFR TKI e.g. gefitinib or erlotinib.
* patients must also have confirmation of tumour T790M mutation status (confirmed positive) after disease progression on the prior EGFR TKI.
* Eastern cooperative oncology group performance status (ECOG PS) of 0-1.
* a minimum life expectancy of 12 weeks.
* At least one lesion, not previously irradiated during the study screening period, that can be accurately measured at baseline according to RECIST 1.1.
* Agree to use routine adequate and effective contraceptive measures during the entire study period and within 6 weeks after the last dose pre-menopausal fertility possible; Female patients need to exclude pregnancy (ie negative pregnancy test) and in non-lactation period.

Exclusion Criteria:

* Treatment with a first or second generation of EGFR-TKI within 10 days of study entry; previous treatment with a third generation of EGFR-TKI.
* Unresolved toxicities from prior therapy.
* Unstable spinal cord compression/brain metastases.
* Severe/uncontrolled systemic diseases, including uncontrolled hypertension, bleeding diatheses or infection.
* QTcF≥470 msec（female）or QTcF≥450 msec（male）during the screening period.
* Severe respiratory diseases such as interstitial lung disease, severe asthma, pulmonary embolism, etc.
* previous treatment with 2 or more lines of Chemotherapy or immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate based on independent radiology review | 24 months
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) as assessed by independent radiology review and investigator | 36 months
  PFS, defined as time from first dose of X-396 to progression or death due to any cause.
Overall survival (OS) | 36 months
  OS, defined as time from first dose of X-396 to death due to any cause.
Duration of response(DoR) | 24 months
  DoR, defined as time from first reponse to disease progression or death
Disease control rate(DCR) | 24 months
  DCR, defined as proportion of complete response, partial response, and disease stabilization to the proportion of patients with evaluable tumors.
Intracranial Progression-free survival(iPFS) | 36 months
  iPFS, defined as the time between baseline brain metastases, from the date of study drug administration to the time between the onset of intracranial tumor progression or death.
Intracranial objective response rate(iORR) | 24 months
  iORR, defined as the proportion of subjects with complete intracranial response, partial intracranial response to subjects with brain metastases at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Study Chair — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu S, Zhang Y, Zhang G, Zhou J, Cang S, Cheng Y, Wu G, Cao P, Lv D, Jian H, Chen C, Jin X, Tian P, Wang K, Jiang G, Chen G, Chen Q, Zhao H, Ding C, Guo R, Sun G, Wang B, Jiang L, Liu Z, Fang J, Yang J, Zhuang W, Liu Y, Zhang J, Pan Y, Chen J, Yu Q, Zhao M, Cui J, Li D, Yi T, Yu Z, Yang Y, Zhang Y, Zhi X, Huang Y, Wu R, Chen L, Zang A, Cao L, Li Q, Li X, Song Y, Wang D, Zhang S, Ding L, Zhang L, Yuan X, Yao L, Shen Z. Efficacy and Safety of Befotertinib (D-0316) in Patients With EGFR T790M-Mutated NSCLC That Had Progressed After Prior EGFR Tyrosine Kinase Inhibitor Therapy: A Phase 2, Multicenter, Single-Arm, Open-Label Study. J Thorac Oncol. 2022 Oct;17(10):1192-1204. doi: 10.1016/j.jtho.2022.06.002. Epub 2022 Jun 18. PMID 35724798